CLINICAL TRIAL: NCT06856655
Title: A Retrospective Data Collection Evaluating Portal Vein Access Sets For Transjugular Intrahepatic Portosystemic Shunt (TIPS) Procedures
Brief Title: Achieving Portal Access With Scorpion Post-Approval Study 2
Acronym: APASS2
Status: Completed | Type: Observational
Sponsor: Argon Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: SCPVA02
Record Dates: First submitted 2025-02-17; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Portal Hypertension; Liver Diseases; Ascites Hepatic; Hydrothorax; Vascular Diseases
Keywords: Transjugular Intrahepatic Portosystemic Shunt; TIPS; Portal Vein Access
MeSH Terms: conditions — Hypertension, Portal; Liver Diseases; Hydrothorax; Vascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Scorpion Portal Vein Access Kit — Procedure/Surgery: Transjugular Intrahepatic Portosystemic Shunt (TIPS)

SUMMARY:
Creation of the parenchymal tract between the portal vein and the hepatic vein is the most difficult and time consuming step in a TIPS procedure. The purpose of this study is to evaluate portal vein access sets during the TIPS procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Scorpion or Scorpion X kit introduced into the vasculature as the initial device for portal vein access

Exclusion Criteria:

1. TIPS procedure was not initiated and/or no portion of the kit was introduced into the vasculature
2. Inaccessible medical records

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The procedure date window for the retrospective data was from 01-Feb-2022 to 05-Feb-2024.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-03-28 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Technical Success | TIPS Procedure
  Creation of the parenchymal tract between the hepatic vein and an intrahepatic branch of the portal vein and confirmed by portogram
Composite of Major Complications | Through 30 days post-TIPS procedure
  Major complications associated with the procedure or study device and defined as complications resulting in an unplanned increase in the level of care, prolonged hospitalization, permanent adverse sequelae, or death.

SECONDARY OUTCOMES:
Number of Participants with Procedural Success | TIPS Procedure
  Successful delivery of the shunt
Device-Related Complications | Through 30 days post-TIPS procedure
  Incidence of complications related to the device as judged by the Investigator

OTHER OUTCOMES:
Portal Vein Access (PVA) Time | TIPS Procedure
  Time (in minutes) from hepatic vein access to portal vein access
Procedure duration | TIPS Procedure
  Interval (in minutes) from first jugular access for TIPS creation to removal of catheters from subject
Fluoroscopy Time | TIPS Procedure
  Measured in minutes
Change in MELD score | up to 30 days post-TIPs procedure
  Change in score from Baseline Characteristics to Follow Up Data
Change in Child-Pugh score | up to 30 days post-TIPs procedure
  Change in score from Baseline Characteristics to Follow Up Data

CONTACTS AND LOCATIONS:
Locations (1):
- Emory University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-09-20): https://cdn.clinicaltrials.gov/large-docs/55/NCT06856655/Prot_SAP_000.pdf